CLINICAL TRIAL: NCT03174873
Title: Laparoscopic Tubal Evaluation in Unexplained Infertility
Brief Title: Tubal Factor in Unexplained Infertility
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohammed Khairy Ali, Lecturer of obstetrics and gynecology, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: TFUI
Record Dates: First submitted 2017-05-29; First posted 2017-06-05 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: Infertility of Tubal Origin
MeSH Terms: interventions — Laparoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Laparoscopy for unexplained infertile couples (Other)
  Interventions: Procedure: laparoscopy

INTERVENTIONS:
Procedure: laparoscopy — Laparoscopy will be done for unexplained infertile couples before starting IVF because not all pathologic lesions that discovered by laparoscope need IVF and so, protect patients from unneeded IVF program

SUMMARY:
Ray and colleagues define "unexplained infertility" as failure to achieve pregnancy when the semen analysis is normal, evidence for ovulation is present, and tubal patency has been established. The efficacy of treatment declines with increasing age and duration of infertility Infertility is a disease , defined by the failure to achieve a successful pregnancy after 12 months or more of appropriate, timed unprotected intercourse or therapeutic donor insemination, barber evaluation and treatment may be justified based on medical history and physical findings and is warranted after 6 months for women over age 35 years.

In unexplained infertility abnormalities are likely to be present but not detected by current methods including semen analysis in the man, assessment of the state of ovulation, ovulation reserve and patency of uterine tubes in the woman.

unexplained infertility is not a rare item of infertility. Approximately 15% of infertility couple will be diagnosed with unexplained infertility after their diagnostic workup Many researches studied the laparoscopic tubal factor like tubo-ovarian relation, tubal kinks and fimbrial pathology. But we need to scope on more tubal factors like fatty mesosalpinx , fimbria ovarica, methylene blue free spill and others

ELIGIBILITY:
Inclusion Criteria:

* women with unexplained infertility.
* women in reproductive period between 20 and 35 years.
* primary or secondary infertility

Exclusion Criteria:

* with age less than 20 years and more than 35 years old
* other causes of infertility other than tubal factor
* Other contraindications for laparoscopy

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2022-04-01 (Actual); Study Completion 2022-10-01 (Actual)

PRIMARY OUTCOMES:
Number of Participants will be diagnosed to have tubal cause of infertility by laparoscopy | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Women Health Hospital - Assiut university, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided